CLINICAL TRIAL: NCT06870851
Title: Machine Learning Based Prediction of Platelet Concentration From ROTEM Measurements
Brief Title: Predicting Platelet Count From Viscoelastic Testing
Status: Active, not recruiting | Type: Observational
Sponsor: Kepler University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: plateletprediction
Record Dates: First submitted 2025-03-03; First posted 2025-03-11 (Actual); Last update posted 2025-03-11 (Actual); Status verified 2025-03

CONDITIONS: Thrombocytopenia
MeSH Terms: conditions — Thrombocytopenia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
Viscoelastic testing is a highly recommended cornerstone of modern coagulation medicine, reducing transfusion needs. A disadvantage of viscoelastic tests is the impossibility of making a definitive statement about the platelet count.

Therefore, the aim of this retrospective observational study is, on the one hand, to predict the platelet count based on standard ROTEM parameters with the help of several machine learning methods and, on the other hand, to detect a low platelet count ( <100000 ml-1 and < 50000 ml-1).

ELIGIBILITY:
Inclusion Criteria:

* ROTEM measurement and platelet count measurement within 3 hours.

Exclusion Criteria:

* under 18 Years
* more than 3 hours between ROTEM and platelet count measurement

Ages: 18 Years to 100 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: surgical patients in the operating room and the intensive care of participating centers
Sampling Method: Non-Probability Sample
Enrollment: 2500 (Estimated)
Dates: Start 2024-10-01 (Actual); Primary Completion 2025-04 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Predicition of platelet conentration from ROTEM measurements using machine learning | Obtained ROTEM analyses are the baseline at all four centres and patients will be included if platelets were determined concomitantly within three hours on the same day.
  Several machine learning techniques for the prediction of the platelet concentration from ROTEM parameters (regression approach), namely linear regression, Random Forest, neural network, gradient boosting machine (GBM) and adaptive boosting (ADA) will be assessed. Describing the quality of these prediction models, the mean square error (MSE), the root of the mean of the square of errors(RMSE), the mean absolute error (MAE), and the root mean squared logarithmic error (RMSLE), and the coefficient of determination (R2) will be used.

CONTACTS AND LOCATIONS:
Locations (1):
- Universitätsklinik für Anästhesie und Intensivmedizin, Linz, Austria